CLINICAL TRIAL: NCT07055971
Title: Development of a Pain Neuroscience Education Intervention to Analyze Conditioned Pain Modulation Mechanisms and the Emotional Processes Underlying Centralized Pain in Patients With Fibromyalgia
Brief Title: Pain Neuroscience Education, Conditioned Pain Modulation and Emotional Processes in Fibromyalgia
Acronym: NEUROPAINFIB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Antonio Casas, Principal Investigator, PhD research and teaching staff of the University of Granada, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUROPAINFIB_2025; 2024/CH/01 (Other Grant/Funding Number: Cátedra Hammam Al Ándalus I+D+I)
Record Dates: First submitted 2025-06-12; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Chronic pain; Health Education; Pain Neuroscience Education; Emotional Intellegence; Condioned Pain Modulation; Central Sensitization
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Health Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuoescience Education (Experimental)
  Interventions: Behavioral: Experimental: Pain Neuoescience Education Group
- Biomedical Education (Active Comparator)
  Interventions: Behavioral: Active Comparator: Biomedical Education Group

INTERVENTIONS:
Behavioral: Experimental: Pain Neuoescience Education Group — The experimental group will receive a pain neuroscience education (PNE) intervention delivered through an in-person, didactic educational model in small groups of 5 to 10 patients. PNE sessions will be conducted once per week for 6 weeks, each lasting approximately 45 to 60 minutes, by a physiotherapist with extensive clinical experience and specialized training in PNE. The content of the sessions will be based on models described in previous studies. Patients will receive detailed information on the neurophysiology and neurobiology of chronic pain and its relationship to fibromyalgia (FM). Pre-prepared PowerPoint presentations will be used to deliver the material in an accessible and engaging manner, employing images, metaphors, anecdotes, and stories to facilitate understanding. All variables will be recorded at baseline (prior to the intervention), at 6 weeks (end of the intervention), at 12 weeks and at 18 weeks.
  Arms: Pain Neuoescience Education
Behavioral: Active Comparator: Biomedical Education Group — The control group will receive two sessions of biomedical education and general guidance on chronic pain and its management, delivered in small groups of 5 to 10 patients with a duration about 45-60 minute. These sessions will also be conducted by the same physiotherapist who delivers the intervention sessions. Both groups will be instructed to continue their usual care and will be encouraged to engage in therapeutic exercise tailored to their physical limitations. All variables will be recorded at baseline (prior to the intervention), at 6 weeks (end of the intervention), at 12 weeks and at 18 weeks
  Arms: Biomedical Education

SUMMARY:
Chronic pain represents a significant public health concern worldwide and is a primary reason why patients seek specialized medical care. Fibromyalgia (FM) is a highly prevalent chronic condition, affecting approximately 2% to 5% of the global population. Its main symptom is widespread, diffuse pain, often accompanied by joint stiffness, persistent fatigue, paresthesia, hyperalgesia, non-restorative sleep, anxiety, cognitive difficulties, and sensory hypersensitivity.

Although the exact pathophysiology of FM remains incompletely understood, alterations in central nervous system (CNS) nociceptive processing are believed to play a fundamental role in the development, propagation, and persistence of pain associated with this condition. Increased sensitivity to both painful and non-painful stimuli-known as central sensitization-may result from changes in neural function and activity, which also impact the emotional and affective regulation of pain perception and experience.

Pain neuroscience education (PNE) is an emerging therapeutic approach that focuses on helping patients reconceptualize and understand their pain through education about the neurophysiology, neuroanatomy, and neurobiology of pain. This intervention aims to promote patient awareness of the origins of their symptoms, reduce hyperactivity within the nervous system, and modify maladaptive beliefs and attitudes related to their pain experience. PNE seeks to enhance patients' capacity to manage emotional, psychological, and environmental factors that influence pain perception-such as beliefs, cultural background, motivation, and body awareness-in order to improve coping strategies in daily activities.

In this study, the investigators aim to analyze the effects of a PNE program on nociceptive processing and emotional-affective modulation in patients with FM. The hypothesis is that the intervention will lead to improvements in markers of nociceptive processing, such as pressure hyperalgesia, conditioned pain modulation (CPM), and temporal summation (TS), all of which are related to descending inhibitory pain pathways. Furthermore, the researchers anticipate enhancements in the emotional and affective mechanisms that underlie centralized pain in this population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia in accordance with the American College of Rheumatology criteria for classifying Fibromyalgia (2016 revision) by a rheumatologist of the Public Health System of Andalusia (Spain)

Exclusion Criteria:

* Presence of liver, cardiac, or renal disease.
* Presence of previous inflammatory rheumatic disease or neurological disorders.
* Presence of infectious processes, fever, hypotension, or respiratory alterations.
* Severe physical disability or severe psychiatric illness.
* Previous surgical intervention prior to the study period.
* Presence of associated comorbidities (chemical hypersensitivity syndrome, chronic fatigue syndrome, interstitial cystitis, etc.).
* Receiving any other non-pharmacological therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Endogenous pain modulation mechanisms_Pressure Pain Hyperalgesia | Six weeks
  Change from baseline in pressure pain hyperalgesia. Pressure pain thresholds (PPTs) will be assessed at the right trapezius and gastrocnemius muscles using a digital algometer. Force will be increased at a rate of 1 kg/s until the participant reports pain. Three measurements will be taken at each site to calculate the mean value.
Endogenous pain modulation mechanisms_Deep Hyperalgesia | Six Weeks
  Change from baseline in deep hyperalgesia. To quantify the level of deep hyperalgesia, the pressure occlusion threshold will be calculated. An occlusion cuff on the left arm will be inflated at 20 mmHg/s until the subject reports pain. After 30 seconds, pain is rated on a verbal numerical rating scale (VNSR) from 0 to 10 to obtain the VNRS1 value. The cuff pressure is then adjusted until the subject reports level 3 pain on the VNRS, obtaining the VNRS3 value.
Endogenous pain modulation mechanisms_ Temporal Summation of pain | Six Weeks
  Change from baseline in the temporal summation (TS) variable of pain, or endogenous pain facilitation. Will be assessed two minutes after the last quantified Pressure pain thresholds (PPT) at both levels (shoulder and calf). Participants will receive 10 pressure pulses perceived as painful, starting at the previously determined mean PPT intensity. Pressure will be increased at a rate of approximately 2 kg/s for each pulse, with 1-second rest intervals between pulses. For each pulse, the pressure will be maintained for 1 second before being released. After the first, fifth, and tenth pulse, participants will be asked to verbally rate their pain on a verbal numerical rating scale (VNRS). The TS measurement variable will be defined as the difference between the VNRS score after the tenth pulse and that after the first pulse
Endogenous pain modulation mechanisms_Conditioned pain modulation | Six Weeks
  change from baseline in Conditioned pain modulation (CPM) or endogenous pain inhibition. To assess CPM, the sequence previously described for the temporal summation of pain will be repeated while a so-called 'heterotopic noxious conditioning stimulus' is applied to the patient. This painful stimulus will consist of placing an occlusion cuff on the left arm. The cuff will be inflated to the pressure previously determined to correspond to a verbal numerical rating scale (VNRS) score of 3, representing a moderate pain intensity stimulus. The CPM measurement variable will be defined as the difference between the initial VNRS score before inflating the cuff and the initial VNRS score during cuff occlusion.

SECONDARY OUTCOMES:
Pain Intensity: Visual Analog Scale | Baseline and 6 weeks
  Change from baseline in pain in the Visual Analog Scale (VAS). Score range between 0-10 cm where 0 is in considerer no pain and 10 is the worst pain
Pain Intensity: Visual Analog Scale | Baseline and 12 weeks
  Change from baseline in pain in the Visual Analog Scale (VAS). Score range between 0-10 cm where 0 is in considerer no pain and 10 is the worst pain
Pain Intensity: Visual Analog Scale | Baseline and 18 weeks
  Change from baseline in pain in the Visual Analog Scale (VAS). Score range between 0-10 cm where 0 is in considerer no pain and 10 is the worst pain
Pressure Pain Threshold | Baseline and 6 weeks
  Change from baseline un pressure pain thresold. A digital pressure algometer will be use to measure the pressure pain thresold bilaterally over the 22 tender points considered by the American College of Rheumatology for Fibromyalgia
Pressure Pain Threshold | Baseline and 12 weeks
  Change from baseline un pressure pain thresold. A digital pressure algometer will be use to measure the pressure pain thresold bilaterally over the 22 tender points considered by the American College of Rheumatology for Fibromyalgia
Pressure Pain Threshold | Baseline and 18 weeks
  Change from baseline un pressure pain thresold. A digital pressure algometer will be use to measure the pressure pain thresold bilaterally over the 22 tender points considered by the American College of Rheumatology for Fibromyalgia
Central Sensitization | Baseline and 6 weeks
  Change from baseline in the Central Sensitization Inventory (CSI). The score ranges from 0 to 100.Higher scores indicate increased frequency and severity of the symptoms
Central Sensitization | Baseline and 12 weeks
  Change from baseline in the Central Sensitization Inventory (CSI). The score ranges from 0 to 100.Higher scores indicate increased frequency and severity of the symptoms
Central Sensitization | Baseline and 18 weeks
  Change from baseline in the Central Sensitization Inventory (CSI). The score ranges from 0 to 100.Higher scores indicate increased frequency and severity of the symptoms
Severity of Fibromyalgia_perceived disability | Baseline and 6 weeks
  Change from baseline in Revised Fibromyalgia Impact Questionnaire (FIQ-R), the score ranges from 0 to 100 . High scores indicate high severity of fibromyalgia symptoms
Severity of Fibromyalgia_perceived disability | Baseline and 12 weeks
  Change from baseline in Revised Fibromyalgia Impact Questionnaire (FIQ-R) , the score ranges from 0 to 100 . High scores indicate high severity of fibromyalgia symptoms
Severity of Fibromyalgia_perceived disability | Baseline and 18 weeks
  Change from baseline in Revised Fibromyalgia Impact Questionnaire (FIQ-R), the score ranges from 0 to 100 . High scores indicate high severity of fibromyalgia symptoms
Fatigue severity | Baseline and 6 weeks
  Change from baseline in the Multidimensional fatigue inventory (MFI) . High scores indicate a greater degree of fatigue
Fatigue severity | Baseline and 12 weeks
  Change from baseline in the Multidimensional fatigue inventory (MFI). High scores indicate a greater degree of fatigue
Fatigue severity | Baseline and 18 weeks
  Change from baseline in the Multidimensional fatigue inventory (MFI). High scores indicate a greater degree of fatigue
Quality of sleep | Baseline and 6 weeks
  Change from baseline in the Pittsburgh Sleep Quality Index (PSQI). The total score varies in a range from 0 to 21 points. Higher scores report poorer sleep quality.
Quality of sleep | Baseline and 12 weeks
  Change from baseline in the Pittsburgh Sleep Quality Index (PSQI). The total score varies in a range from 0 to 21 points. Higher scores report poorer sleep quality.
Quality of sleep | Baseline and 18 weeks
  Change from baseline in the Pittsburgh Sleep Quality Index (PSQI). The total score varies in a range from 0 to 21 points. Higher scores report poorer sleep quality.
Psychological aspects and common symptoms of anxiety | Baseline and 6 weeks
  Change from baseline in the Beck Anxiety Inventory (BAI). Total score range from 0 to 63 points, with high scores indicating a higher degree of anxiety
Psychological aspects and common symptoms of anxiety | Baseline and 12 weeks
  Change from baseline in the Beck Anxiety Inventory (BAI). Total score range from 0 to 63 points, with high scores indicating a higher degree of anxiety
Psychological aspects and common symptoms of anxiety | Baseline and 18 weeks
  Change from baseline in the Beck Anxiety Inventory (BAI). Total score range from 0 to 63 points, with high scores indicating a higher degree of anxiety
Fear of movement_ Kinesiophobia | Baseline and 6 weeks
  Change from baseline in Tampa Scale of Kinesiophobia (TSK). The total score ranges from 11 to 44 points, with higher scores indicating greater levels of kinesiophobia
Fear of movement_ Kinesiophobia | Baseline and 12 weeks
  Change from baseline in Tampa Scale of Kinesiophobia (TSK). The total score ranges from 11 to 44 points, with higher scores indicating greater levels of kinesiophobia
Fear of movement_ Kinesiophobia | Baseline and 18 weeks
  Change from baseline in Tampa Scale of Kinesiophobia (TSK). The total score ranges from 11 to 44 points, with higher scores indicating greater levels of kinesiophobia
Pain Catastrophizing | Baseline and 6 weeks
  Change from baseline in the Pain Catastrophizing Scale (PCS). Score range is from 0 to 52; higher scores indicate a greater frequency of catastrophic thoughts
Pain Catastrophizing | Baseline and 12 weeks
  Change from baseline in the Pain Catastrophizing Scale (PCS). Score range is from 0 to 52; higher scores indicate a greater frequency of catastrophic thoughts
Pain Catastrophizing | Baseline and 18 weeks
  Change from baseline in the Pain Catastrophizing Scale (PCS). Score range is from 0 to 52; higher scores indicate a greater frequency of catastrophic thoughts
Perceived Emotional Intelligence | Baseline and 6 weeks
  Change from baseline in Trait Meta-Mood Scale (TMMS-24) This scale consists of 24 items distributed across 3 subscales that assess emotional attention, emotional clarity, and emotional repair. Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Normal scores are considered to range from 22 to 35 points for the emotional attention dimension, and from 24 to 35 points for the emotional clarity and emotional repair dimensions
Perceived Emotional Intelligence | Baseline and 12 weeks
  Change from baseline in Trait Meta-Mood Scale (TMMS-24) This scale consists of 24 items distributed across 3 subscales that assess emotional attention, emotional clarity, and emotional repair. Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Normal scores are considered to range from 22 to 35 points for the emotional attention dimension, and from 24 to 35 points for the emotional clarity and emotional repair dimensions
Perceived Emotional Intelligence | Baseline and 18 weeks
  Change from baseline in Trait Meta-Mood Scale (TMMS-24) This scale consists of 24 items distributed across 3 subscales that assess emotional attention, emotional clarity, and emotional repair. Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Normal scores are considered to range from 22 to 35 points for the emotional attention dimension, and from 24 to 35 points for the emotional clarity and emotional repair dimensions
Global Level of Empathy | Baseline and 6 weeks
  Change from baseline in the Interpersonal Reactivity Index (IRI). This scale consists of 28 items that assess both the cognitive aspect and the emotional response of the individual when adopting an empathetic attitude. Each item is rated on a Likert scale ranging from 0 (does not describe me well) to 4 (describes me very well)
Global Level of Empathy | Baseline and 12 weeks
  Change from baseline in the Interpersonal Reactivity Index (IRI). This scale consists of 28 items that assess both the cognitive aspect and the emotional response of the individual when adopting an empathetic attitude. Each item is rated on a Likert scale ranging from 0 (does not describe me well) to 4 (describes me very well)
Global Level of Empathy | Baseline and 18 weeks
  Change from baseline in the Interpersonal Reactivity Index (IRI). This scale consists of 28 items that assess both the cognitive aspect and the emotional response of the individual when adopting an empathetic attitude. Each item is rated on a Likert scale ranging from 0 (does not describe me well) to 4 (describes me very well)
Cognitive and Affective Levels of Empathy | Baseline and 6 weeks
  Change from baseline in Cognitive and Affective Empathy Test (TECA) It consists of 33 items distributed across 4 subscales . Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater levels of empathy
Cognitive and Affective Levels of Empathy | Baseline and 12 weeks
  Change from baseline in Cognitive and Affective Empathy Test (TECA) It consists of 33 items distributed across 4 subscales . Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater levels of empathy
Cognitive and Affective Levels of Empathy | Baseline and 18 weeks
  Change from baseline in Cognitive and Affective Empathy Test (TECA) It consists of 33 items distributed across 4 subscales . Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater levels of empathy
Positive and Negative Affect of Emotions and Feelings | Baseline and 6 weeks
  Change from baseline in Positive and Negative Affect Schedule (PANAS). It consists of 20 items distributed across two subscales that assess various emotions and feelings of a positive or negative nature. Each item is rated on a Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely). The total score ranges from 10 to 50 points, with higher scores indicating a greater presence of the specific type of affectTime
Positive and Negative Affect of Emotions and Feelings | Baseline and 12 weeks
  Change from baseline in Positive and Negative Affect Schedule (PANAS). It consists of 20 items distributed across two subscales that assess various emotions and feelings of a positive or negative nature. Each item is rated on a Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely). The total score ranges from 10 to 50 points, with higher scores indicating a greater presence of the specific type of affectTime
Positive and Negative Affect of Emotions and Feelings | Baseline and 18 weeks
  Change from baseline in Positive and Negative Affect Schedule (PANAS). It consists of 20 items distributed across two subscales that assess various emotions and feelings of a positive or negative nature. Each item is rated on a Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely). The total score ranges from 10 to 50 points, with higher scores indicating a greater presence of the specific type of affectTime
Emotional Well-being | Baseline and 6 weeks
  Change from baseline in the Mental Health-5 (MH-5) Scale It consists in a subscale of the Short Form-36 Health Survey, with 5 items related to the area of emotional well-being and assesses the mental health of the participants. Each item is rated on a Likert scale ranging from 1 (always) to 6 (never). Higher scores are associated with better mental health
Emotional Well-being | Baseline and 12 weeks
  Change from baseline in the Mental Health-5 (MH-5) Scale It consists in a subscale of the Short Form-36 Health Survey, with 5 items related to the area of emotional well-being and assesses the mental health of the participants. Each item is rated on a Likert scale ranging from 1 (always) to 6 (never). Higher scores are associated with better mental health
Emotional Well-being | Baseline and 18 weeks
  Change from baseline in the Mental Health-5 (MH-5) Scale It consists in a subscale of the Short Form-36 Health Survey, with 5 items related to the area of emotional well-being and assesses the mental health of the participants. Each item is rated on a Likert scale ranging from 1 (always) to 6 (never). Higher scores are associated with better mental health
Patients' knowledge levels regarding the neurophysiology of pain | Baseline and 6 weeks
  Change from baseline in the Revised Neurophysiology of Pain Questionnaire (R-NPQ). The questionnaire consists of 13 statements about pain (True/False/Don't know), with a total score ranging from 0 to 13 (sum of all correct items).
Patients' knowledge levels regarding the neurophysiology of pain | Baseline and 12 weeks
  Change from baseline in the Revised Neurophysiology of Pain Questionnaire (R-NPQ). The questionnaire consists of 13 statements about pain (True/False/Don't know), with a total score ranging from 0 to 13 (sum of all correct items).
Patients' knowledge levels regarding the neurophysiology of pain | Baseline and 18 weeks
  Change from baseline in the Revised Neurophysiology of Pain Questionnaire (R-NPQ). The questionnaire consists of 13 statements about pain (True/False/Don't know), with a total score ranging from 0 to 13 (sum of all correct items).
Pain vigilance and awareness | Baseline and 6 weeks
  Change from baseline in the 9-item short form of the Pain Vigilance and Awareness Questionnaire (PVAQ-9). Each item is rated on a Likert scale from 0 (never) to 5 (always), with a total score ranging from 0 to 45 points. The optimal cutoff point for identifying women with fibromyalgia who experience poorer daily functioning is set at 24.5 points
Pain vigilance and awareness | Baseline and 12 weeks
  Change from baseline in the 9-item short form of the Pain Vigilance and Awareness Questionnaire (PVAQ-9). Each item is rated on a Likert scale from 0 (never) to 5 (always), with a total score ranging from 0 to 45 points. The optimal cutoff point for identifying women with fibromyalgia who experience poorer daily functioning is set at 24.5 points
Pain vigilance and awareness | Baseline and 18 weeks
  Change from baseline in the 9-item short form of the Pain Vigilance and Awareness Questionnaire (PVAQ-9). Each item is rated on a Likert scale from 0 (never) to 5 (always), with a total score ranging from 0 to 45 points. The optimal cutoff point for identifying women with fibromyalgia who experience poorer daily functioning is set at 24.5 points

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Casas Barragán, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No